CLINICAL TRIAL: NCT01209728
Title: A Randomized Clinical Trial to Study the Effects of Simulated Driving on Primary Insomniacs
Brief Title: Effects of Insomnia on Simulated Driving (MK-0000-183-00)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0000-183
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Insomnia
Keywords: insomnia; insomniacs; simulated driving; alcohol; ethanol
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary insomnia patients and healthy subjects (Experimental): Elderly participants, including primary insomnia patients and healthy subjects
  Interventions: Other: Placebo/ethanol (blinded)

INTERVENTIONS:
Other: Placebo/ethanol (blinded) — Elderly participants, including primary insomnia patients and healthy subjects will be administered i.v. ethanol or placebo in a blinded manner
  Other Names: Placebo or ethanol (blinded)

SUMMARY:
This is a double-blind, parallel design study in elderly primary insomnia patients and demographically matched controls. The objectives if this study are primarily: 1. To determine if functional deficits in simulated driving performance can be demonstrated in primary insomnia patients, and detected in healthy volunteers, impaired by alcohol; and secondarily: 2. To compare simulated driving performance deficits in elderly primary insomnia patients to those in healthy elderly volunteers impaired by alcohol, for at least one of the following driving endpoints: standard deviation of lane position (SDLP), standard deviation of speed (speed deviation), lane excursions, and a driving composite score.

ELIGIBILITY:
Inclusion Criteria A patient or subject may participate in the study if, at least, the ALL of the criteria below are met.

The participant:

* Is a male or female of non-childbearing potential and 65 years of age or older at prestudy (screening);
* Has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months prior to screening;
* Has a current valid driver's license;
* Their regular bedtime is between 9 pm (21:00) and 12 am (00:00);
* During the study, are willing to refrain from napping;

Additionally, a primary insomnia patient must meet the following inclusion criteria:

* Has a diagnosis of Primary Insomnia;
* Reports total sleep time of < 6 hours on at least 3 out of 7 nights each week during the 4 weeks prior to screening;
* Reports spending 6 to 9 hours nightly in bed on at least 3 out of 7 nights each week during the 4 weeks prior to screening.

Exclusion Criteria :

A patient may not participate in the study if ANY of the criteria below (among others determined by the study staff) apply.

The participant:

* Has visual or auditory impairment;
* Has a history of clinically significant endocrine (including diabetes), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases;
* Has a history of neoplastic disease ;
* Is taking, or plans to take, one or more of the following medications (non-inclusive), within the 2 weeks prior to screening and throughout the course of the study: Centrally acting anticholinergics or antihistamines; Melatonin; Anticonvulsants; Antipsychotics; Anxiolytics; Benzodiazepines; Hypnotics; Any CNS depressants; Over-the-counter medications that could affect sleep; Stimulants; Diet pills; Anti-depressants; Disulfiram;
* Has a positive screening urine drug test (e.g., positive for benzodiazepines, cannabinoids, cocaine, etc.);
* Has a lifetime history of bipolar disorder, a psychotic disorder, or posttraumatic stress disorder or a psychiatric condition requiring treatment with a prohibited medication; or other current psychiatric condition that, in the investigator's opinion, would interfere with the subject/patient's ability to participate in the study ;
* Has evidence of suicidality;
* Has a history of transmeridian travel (across > 3 time zones or > 3 hour time difference) within two weeks prior to screening or anticipates transmeridian travel during the study;
* Has a history of shift work (defined as permanent night shift or rotating day/night shift work) within the past two weeks prior to screening or anticipates need to perform shift work during the study;
* Has a history or diagnosis of any of following conditions, in the opinion of the investigator: Narcolepsy; Cataplexy (familial or idiopathic); Circadian Rhythm Sleep Disorder; Parasomnia including nightmare disorder, sleep terror disorder, sleepwalking disorder, and REM behavior disorder; Sleep-related Breathing Disorder (obstructive or central sleep apnea syndrome, central alveolar hypoventilation syndrome); Periodic Limb Movement Disorder; Restless Legs Syndrome; Primary Hypersomia; Excessive Daytime Sleepiness (EDS), not attributable to Primary Insomnia
* Has a recent and/or active history of a confounding neurological disorder, including but not limited to: seizure disorder, stroke, transient ischemic attack, multiple sclerosis, cognitive impairment, or significant head trauma with sustained loss of consciousness and residual impairment within the last 10 years;
* Has a history of allergy, exceptional sensitivity, or adverse reaction to alcohol;
* Has a significant history of motion sickness or demonstrates significant simulator sickness during practice drives at screening;
* Consumes excessive amounts of alcohol or subject or patient consumes alcohol to promote sleep (i.e., within 3 hours before going to bed);
* Has never consumed alcohol;
* Consumes excessive amounts of coffee, tea, cola, or other caffeinated beverages.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

PRIMARY OUTCOMES:
Simulated driving variables | Evaluated on, up to, 3 different days, with 2 driving sessions of ~65 minutes each day.
  Simulated driving variables which may include (standard deviation of lane position (SDLP), speed deviation, lane excursions, or a composite score of several driving variables).

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Simen AA, Gargano C, Cha JH, Drexel M, Bautmans A, Heirman I, Laethem T, Hochadel T, Gheyle L, Bleys K, Beals C, Stoch A, Kay GG, Struyk A. A randomized, crossover, placebo-controlled clinical trial to assess the sensitivity of the CRCDS Mini-Sim to the next-day residual effects of zopiclone. Ther Adv Drug Saf. 2015 Jun;6(3):86-97. doi: 10.1177/2042098615579314. PMID 26240742